CLINICAL TRIAL: NCT00702897
Title: Ambulatory Surgery of Lower Extremity Varicose Vein
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Far Eastern Memorial Hospital, Far Eastern Memorial Hospital
Other Study IDs: FEMH-96041
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
OBJECTIVE: To retrospectively analyze the results of ambulatory treatment on Taiwanese patients with primary varicosities of the lower extremities including the use of endovenous laser, phlebectomy, and sclerotherapy.

METHODS: We routinely used tumescent anesthesia and ultrasound-guided approaches for the application of endovenous laser. Vein access was achieved by either a percutaneous or stab wound. The laser power was usually 10 - 20 watts; laser treatment usually was begun from 4-10 cm below the saphenofemoral junction, and stopped around the knee, not over 10 cm below the knee. In the same operation, we used Mueller's phlebectomy and/or sclerotherapy if there were prominent branch varicosities. We instructed each patient to walk around immediately after the operation, to go home, and to come back 1-3 days later for follow-up. Ultrasound scan and venous function follow-up was scheduled at 1 month, 6 months, 12 months, and then annually.

ELIGIBILITY:
Inclusion Criteria:

* All patients with varicose veins who underwent endovenous laser treatment for GSV reflux in our hospital were reviewed

Exclusion Criteria:

* poor general health, inability to walk, active inflammation of varicose veins, deep venous occlusion disease, hypercoagulability, pregnancy and breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with varicose veins who underwent endovenous laser treatment for GSV reflux in our hospital were reviewed.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-01

CONTACTS AND LOCATIONS:
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan